CLINICAL TRIAL: NCT06533514
Title: Rapid Diagnosis of Severe Respiratory Tract Infectious Diseases and Screening of Biomarkers for Stratified Diagnosis
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Deputy chief physician, Chinese PLA General Hospital
Other Study IDs: Pneumonia and Biomarkers
Record Dates: First submitted 2024-07-23; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Severe Pneumonia; Biomarkers
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild: According to the APACHE II score, SOFA score and PSI score, the enrolled patients were divided into three groups: mild, moderate and severe.
- moderate: According to the APACHE II score, SOFA score and PSI score, the enrolled patients were divided into three groups: mild, moderate and severe.
- severe: According to the APACHE II score, SOFA score and PSI score, the enrolled patients were divided into three groups: mild, moderate and severe.

SUMMARY:
The purpose of this study is to clarify the biomarkers for rapid diagnosis and stratified diagnosis of severe respiratory tract infectious diseases through clinical experiments.

DETAILED DESCRIPTION:
Methods: The relationship between relevant biomarkers and stratified diagnosis was analyzed by collecting laboratory and etiological examinations of patients with severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for severe pneumonia；
* Age≥18 years old and < 80 years old；
* Willing to sign informed consent for the course of the study；

Exclusion Criteria:

* Patients with intracranial hypertension, acute coronary syndrome, pleural fistula, pneumothorax, or subcutaneous emphysema;
* Pregnant and lactating patients;
* Severely hemodynamically unstable (an increase in vasopressors by more than 30% in the first 6 hours, or norepinephrine >0.5mg/kg/min);
* Those who do not consent to participate in this study；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Meets the diagnostic criteria for severe pneumonia；
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The relationship between the patient's specific biomarker levels and clinical outcomes. | 1 mounth
  Treatment failure rate, Mortality rates, SOFA rating scale

IPD SHARING:
Plan to Share IPD: No